CLINICAL TRIAL: NCT01662167
Title: Comparison of Single and Multiple-dose Methotrexate Therapy for Ectopic Pregnancy: a Clinical Trail
Brief Title: Comparison of Single and Multiple-dose Methotrexate Therapy for Ectopic Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad E Shahrzad, MD, Dr, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1133-3069
Record Dates: First submitted 2012-08-05; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy, Ectopic
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Single Person

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Multiple dose mtx (Experimental): mtx
  Interventions: Drug: Multipe
- Single Dose (Experimental): In the single dose regimen, 50 mg/m2 intramuscular methotrexate was given on day one and hCG level was measured on days four and seven. If the hCG level did not decrease by 15% between day four and seven, a second dose of methotrexate was injected on day seven, hCG level was measured weekly until a level of 15 mlU/ml or less was achieved
  Interventions: Drug: Single

INTERVENTIONS:
Drug: Single — In the single dose regimen, 50 mg/m2 intramuscular methotrexate was given on day one and hCG level was measured on days four and seven. If the hCG level did not decrease by 15% between day four and seven, a second dose of methotrexate was injected on day seven, hCG level was measured weekly until a level of 15 mlU/ml or less was achieved
  Arms: Single Dose
Drug: Multipe — In the multiple dose regimen, 1 mg/kg/day intramuscular methotrexate was given on days one, three, five and seven and 0.1 mg/kg/day intramuscular Citrovoram factor was administered on days two, four, six and eight until serum hCG level decreased 15% in 48 hours or four doses of methotrexate was given weekly until serum hCG level of 15 mlU/ml or less was obtained
  Arms: Multiple dose mtx

SUMMARY:
The aim of this study was to compare single dose Methotrexate (MTX) to multiple dose MTX.

ELIGIBILITY:
Inclusion Criteria:

* unruptured tubal EP
* gestational mass of less than or equal to 3.5 cm in ultrasonography report

Exclusion Criteria:

* hemodynamic instability
* contraindications related to the use of MTX
* hepatic
* renal and active pulmonary diseases
* peptic ulcer
* immune deficiency status
* alcohol abuse
* blood dyscreasia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
hCG level decrease | 4 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Shariaty Hospital, Bandar Abbas, Hormozgan, Iran